CLINICAL TRIAL: NCT01565083
Title: A Two-cohort, Open-label, Multicenter Phase II Trial Assessing the Efficacy and Safety of Pertuzumab Given in Combination With Trastuzumab and Vinorelbine in First Line Patients With HER2-positive Advanced (Metastatic or Locally Advanced) Breast Cancer
Brief Title: A Study to Assess Efficacy and Safety of Pertuzumab Given in Combination With Trastuzumab and Vinorelbine in Participants With Metastatic or Locally Advanced Human Epidermal Growth Factor Receptor (HER) 2-Positive Breast Cancer
Acronym: VELVET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO27782; 2011-003308-18 (EudraCT Number)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab; Vinorelbine

ARMS (2):
- Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion (Experimental): Pertuzumab will be administered as IV infusion on Day 1 of the first treatment cycle (1 cycle = 21 days) as a loading dose of 840 milligrams (mg), followed by 420 mg on Day 1 of each subsequent cycle. Trastuzumab will be administered as IV infusion on Day 2 of the first treatment cycle as a loading dose of 8 mg per kilogram (mg/kg), followed by 6 mg/kg on Day 2 of each subsequent cycle. Vinorelbine IV infusion (will be administered after trastuzumab) on Day 2 and Day 9 of the first treatment cycle at a dose of 25 mg per meter-squared (mg/m^2) followed by 30-35 mg/m^2 on Day 2 and Day 9 of each subsequent cycle. Pertuzumab and trastuzumab will be administered sequentially in separate infusion bags, followed by vinorelbine until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end (up to 47 cycles).
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Vinorelbine
- Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion (Experimental): Pertuzumab will be administered as IV infusion on Day 1 of the first treatment cycle as a loading dose of 840 mg, followed by 420 mg on Day 1 of each subsequent cycle. Trastuzumab will be administered as IV infusion on Day 2 of the first treatment cycle as a loading dose of 8 mg/kg, followed by 6 mg/kg on Day 1 of each subsequent cycle. Vinorelbine IV infusion on Day 2 and Day 9 of the first treatment cycle at a dose of 25 mg/m^2 followed by 30-35 mg/m^2 on Day 1 and Day 8 of each subsequent cycle. If administration of all 3 drugs is well tolerated in Cycle 1, then on Day 1 of each subsequent cycle, pertuzumab 420 mg and trastuzumab 6 mg/kg will be administered in a single infusion bag, followed by vinorelbine until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end (up to 47 cycles).
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pertuzumab — Loading dose of 840 mg on Day 1 of first 21-day cycle, followed by 420 mg on Day 1 of each subsequent cycle.
  Other Names: Perjeta
Drug: Trastuzumab — Loading dose of 8 mg/kg on Day 1 of first 21-day cycle, followed by 6 mg/kg on Day 1 or 2 of each subsequent cycle.
  Other Names: Herceptin
Drug: Vinorelbine — A dose of 25 mg/m^2 followed by 30-35 mg/m^2 on Days 2 and 9 of the first 21-day cycle and on Days 1 and 8 (or Days 2 and 9) of each subsequent cycle.

SUMMARY:
This two-cohort, open-label, multicenter, phase 2 study will assess the safety and efficacy of pertuzumab given in combination with trastuzumab (Herceptin) and vinorelbine in first line participants with metastatic or locally advanced HER2-positive breast cancer. Participants will receive pertuzumab and trastuzumab administered sequentially as separate intravenous (IV) infusions (followed by vinorelbine) and conventional sequential administration of pertuzumab and trastuzumab in separate infusion bags, followed by vinorelbine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed and documented adenocarcinoma of the breast with metastatic or locally advanced disease not amenable to curative resection
* HER2-positive as assessed by local laboratory on primary or metastatic tumor
* At least one measurable lesion and/or non-measurable disease evaluable according to RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Left ventricular ejection fraction (LVEF) of at least 55%
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Previous systemic non-hormonal anti-cancer therapy in the metastatic or locally advanced breast cancer setting
* Previous approved or investigative anti-HER2 agents in any breast cancer treatment setting, except trastuzumab and/or lapatinib in the adjuvant or neoadjuvant setting
* Disease progression while receiving trastuzumab and/or lapatinib in the adjuvant or neoadjuvant setting
* Disease-free interval from completion of adjuvant or neoadjuvant systemic non-hormonal treatment to recurrent disease of less than 6 months
* History of persistent Grade 2 or higher (National Cancer Institute Common Terminology Criteria [NCI-CTC], Version 4.0) hematological toxicity resulting from previous adjuvant or neoadjuvant therapy
* Radiographic evidence of central nervous system metastases that are not well controlled with local therapy (irradiation or surgery)
* Current peripheral neuropathy of NCI-CTC, version 4.0 Grade 3 or greater
* History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, or cancers with a similar curative outcome as those mentioned above
* Serious uncontrolled concomitant disease that would contraindicate the use of any of the investigational drugs used in this study or would put the participants at high risk for treatment-related complications
* Inadequate hematologic, liver, or renal function
* Uncontrolled hypertension or clinically significant cardiovascular disease
* Hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection
* Current chronic daily treatment with corticosteroids (>/= 10 mg/day methylprednisolone or equivalent), excluding inhaled steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (75):
- United States (16):
  - Tucson, Arizona
  - Stanford, California
  - Denver, Colorado
  - Hollywood, Florida
  - Miami, Florida
  - Plantation, Florida
  - Marietta, Georgia
  - Boston, Massachusetts
  - Morristown, New Jersey
  - Durham, North Carolina
  - Columbus, Ohio
  - Houston, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Fredericksburg, Virginia
  - Seattle, Washington
- Brazil (3):
  - Rio de Janeiro, Rio de Janeiro
  - Barretos, São Paulo
  - São Paulo, São Paulo
- Denmark (4):
  - Herlev
  - Herning
  - København Ø
  - Odense
- France (13):
  - Avignon
  - Bobigny
  - Caen
  - La Tronche
  - Mont-de-Marsan
  - Paris
  - Périgueux
  - Pierre-Bénite
  - Plérin
  - Rouen
  - Strasbourg
  - Tours
  - Villejuif
- Germany (19):
  - Cologne
  - Dortmund
  - Dresden
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Georgsmarienhütte
  - Goslar
  - Gütersloh
  - Hamburg
  - Heidelberg
  - Kaiserslautern
  - Kassel
  - Lebach
  - Leer
  - Moers
  - München
  - Neumarkt
  - Ravensburg
  - Würselen
- Italy (10):
  - Bologna, Emilia-Romagna
  - Aviano, Friuli Venezia Giulia
  - Rome, Lazio
  - Genoa, Liguria
  - Cremona, Lombardy
  - Monza, Lombardy
  - Lido di Camaiore, Tuscany
  - Pisa, Tuscany
  - Terni, Umbria
  - Negrar, Veneto
- Spain (10):
  - Badajoz, Badajoz
  - Palma de Mallorca, Balearic Islands
  - Terrassa, Barcelona
  - Santander, Cantabria
  - Barbastro, Huesca
  - Madrid, Madrid
  - Málaga, Malaga
  - Oviedo, Principality of Asturias
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia

REFERENCES:
- [Derived] Perez EA, Lopez-Vega JM, Petit T, Zamagni C, Easton V, Kamber J, Restuccia E, Andersson M. Safety and efficacy of vinorelbine in combination with pertuzumab and trastuzumab for first-line treatment of patients with HER2-positive locally advanced or metastatic breast cancer: VELVET Cohort 1 final results. Breast Cancer Res. 2016 Dec 13;18(1):126. doi: 10.1186/s13058-016-0773-6. PMID 27955684

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to non-randomized nature of the study (single infusion cohort started enrollment only after separate infusion cohort recruitment was completed) and different baseline characteristics of participants, the comparison between the 2 cohorts was not performed. Hence, the efficacy and safety results for the 2 cohorts should be considered separately.
Groups:
- Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion: Pertuzumab intravenous (IV) infusion at a loading dose of 840 milligrams (mg) on Day 1 of Cycle 1 (cycle length = 21 days), followed by 420 mg on Day 1 of each subsequent cycle. Trastuzumab IV infusion at a loading dose of 8 mg per kilogram (mg/kg) on Day 2 of Cycle 1, followed by 6 mg/kg on Day 2 of each subsequent cycle. Vinorelbine IV infusion (administered after trastuzumab) at a dose of 25 mg per meter-squared (mg/m^2) on Day 2 and Day 9 of Cycle 1, followed by 30-35 mg/m^2 on Day 2 and Day 9 of each subsequent cycle. Pertuzumab and trastuzumab were administered sequentially in separate infusion bags, followed by vinorelbine until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end (up to 47 cycles).
- Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion: Pertuzumab IV infusion at a loading dose of 840 mg on Day 1 of Cycle 1 (cycle length = 21 days), followed by 420 mg on Day 1 of each subsequent cycle. Trastuzumab IV infusion at a loading dose of 8 mg/kg on Day 2 of Cycle 1, followed by 6 mg/kg on Day 1 of each subsequent cycle. Vinorelbine IV infusion at a dose of 25 mg/m^2 on Day 2 and Day 9 of Cycle 1, followed by 30-35 mg/m^2 on Day 1 and Day 8 of each subsequent cycle. If administration of all 3 drugs was well tolerated in Cycle 1, then on Day 1 of each subsequent cycle, pertuzumab 420 mg and trastuzumab 6 mg/kg was administered in a single infusion bag, followed by vinorelbine until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end (up to 47 cycles).
Period: Overall Study
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Started | 106 | 107
Completed | 73 | 68
Not Completed | 33 | 39
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 2 | 7
Not completed — Death | 22 | 23
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled into the study.
Groups:
- Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion: Pertuzumab IV infusion at a loading dose of 840 mg on Day 1 of Cycle 1 (cycle length = 21 days), followed by 420 mg on Day 1 of each subsequent cycle. Trastuzumab IV infusion at a loading dose of 8 mg/kg on Day 2 of Cycle 1, followed by 6 mg/kg on Day 2 of each subsequent cycle. Vinorelbine IV infusion (administered after trastuzumab) at a dose of 25 mg/m^2 on Day 2 and Day 9 of Cycle 1, followed by 30-35 mg/m^2 on Day 2 and Day 9 of each subsequent cycle. Pertuzumab and trastuzumab were administered sequentially in separate infusion bags, followed by vinorelbine until disease progression, unacceptable toxicity, withdrawal of consent, death, or predefined study end (up to 47 cycles).
- Total: Total of all reporting groups
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion | Total
Number analyzed (Participants) | 106 | 107 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (11.80) | 55.6 (13.17) | 56.2 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 106 | 212
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response (BOR) as Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Tumor response was assessed by investigator according to RECIST v1.1. BOR was defined as percentage of participants with a confirmed complete response (CR) or partial response (PR). All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total or pathological nodes (with short axis [SA] of at least (>/=) 15 millimeter [mm]) were identified as target lesions (TLs) and measured and recorded at baseline. A sum of diameters (longest for non-nodal lesions, SA for nodal lesions) for all TLs was calculated and reported as baseline sum of diameters (SD). All other lesions (or sites of disease) were identified as non-TLs. CR: disappearance of all TLs and SA reduction to less than (<) 10 mm for nodal TLs/ non-TLs. PR: >/=30 percent (%) decrease in SD of TLs, taking as reference baseline SD. Confirmation of response at 2 consecutive tumor assessments >/=4 weeks apart was required. The 95% confidence interval (CI) was computed using Clopper-Pearson approach.
Time Frame: Baseline, every 3 cycles up to 36 months, and every 6 cycles thereafter if progression free after 36 months, 28 days after end of treatment, every 3 months thereafter (maximum up to approximately 3.5 years)
Population: ITT population. Only participants with measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 89 | 91
percentage of participants | 74.2 [63.8 to 82.9] | 63.7 [53.0 to 73.6]

2. Secondary Outcome: Time to Response as Assessed by Investigator According to RECIST v 1.1
Description: For participants with a BOR of CR or PR, time to response = (Date of first confirmed CR/PR - Date of first study treatment) + 1. For participants without a CR or PR, time to response = (Date of adequate last tumor assessment - Date of first study treatment) + 1. For participant with no tumor assessment (or if all assessments were progressive disease [PD]) the censoring day was set to date of first study treatment +1. CR: the disappearance of all TLs and SA reduction to <10 mm for nodal TLs/ non-TLs. PR: >/=30% decrease in SD of TLs, taking as reference the baseline SD. Confirmation of response at 2 consecutive tumor assessments >/=4 weeks apart was required. PD: >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. The 95% CI was computed using log-log transformation.
Time Frame: as for outcome 1
Population: ITT population. Only participants with measurable disease at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 89 | 91
months | 2.1 [2.0 to 2.2] | 2.2 [2.1 to 4.4]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator According to RECIST v 1.1
Description: DOR, in participants with a BOR of CR or PR, was defined as the period from the date of initial PR or CR until the date of PD or death from any cause. Participants with no documented PD or death after CR or PR were censored at the last date at which they were known to have had the CR or PR, respectively (regardless of the response at intermediate assessments). CR: the disappearance of all TLs and SA reduction to <10 mm for nodal TLs/ non-TLs. PR: >/=30% decrease in SD of TLs, taking as reference the baseline SD. Confirmation of response at 2 consecutive tumor assessments >/=4 weeks apart was required. PD: >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. The 95% CI was computed using log-log transformation.
Time Frame: as for outcome 1
Population: ITT population. Only participants with a BOR of CR or PR and with measurable disease at baseline were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 66 | 58
months | 13.3 [10.6 to 16.2] | 11.8 [7.5 to 17.9]

4. Secondary Outcome: Percentage of Participants With Disease Progression as Assessed by Investigator According to RECIST v1.1 or Death From Any Cause
Description: PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. Percentage of participants with radio-graphically documented PD as assessed by investigator according to RECIST v1.1 or death due to any cause was reported.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
percentage of participants | 69.8 | 67.3

5. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Investigator According to RECIST v 1.1
Description: PFS was defined as the time from first intake of any study medication until the first radio-graphically documented PD as assessed by investigator according to RECIST v1.1 or death due to any cause, whichever occurred first. Participants with no PFS events were censored at the time of the last evaluable tumor assessment. Participants with no baseline or no tumor assessment after the baseline visit were censored on the date of first study treatment. PD: >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. Participants who had radio-graphically documented PD as assessed by investigator according to RECIST v1.1 or died due to any cause were considered as having an event. The median PFS was estimated using Kaplan-Meier method. The 95% CI was computed using log-log transformation.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
months | 14.3 [11.2 to 17.5] | 11.5 [10.3 to 15.8]

6. Secondary Outcome: Percentage of Participants With Disease Progression as Assessed by Investigator According to RECIST v1.1
Description: PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. Percentage of participants with radio-graphically documented PD as assessed by investigator according to RECIST v1.1 was reported.
Time Frame: as for outcome 1
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
percentage of participants | 67.9 | 61.7

7. Secondary Outcome: Time to Progression (TTP) as Assessed by Investigator According to RECIST v 1.1
Description: TTP was defined as the time from first intake of any study medication until the first radio-graphically documented PD as assessed by investigator according to RECIST v1.1. Participants who did not have a radio-graphically documented PD and had died due to reason other than PD were censored on the last available tumor assessment prior to the death date. Participants with no baseline or no tumor assessment after the baseline visit were censored on the date of first study treatment. PD was defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. Participants who had radio-graphically documented PD as assessed by investigator according to RECIST v1.1 were considered as having an event. The median TTP was estimated using Kaplan-Meier method. The 95% CI was computed using log-log transformation.
Time Frame: as for outcome 1
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
months | 14.9 [11.3 to 17.9] | 12.8 [10.4 to 17.1]

8. Secondary Outcome: Percentage of Participants Who Died From Any Cause
Description: Percentage of participants who died due to any cause was reported.
Time Frame: Baseline until death (up to approximately 3.5 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
percentage of participants | 21.7 | 21.5

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first intake of any study medication to the date of death, regardless of the cause of death. Participants who were known to be alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study treatment, and participants with no post-baseline information were censored at the date of first study treatment plus 1 day. Participants who died due to any cause were considered as having an event. The median OS was estimated using Kaplan-Meier method. The 95% CI was computed using log-log transformation.
Time Frame: Baseline until death (up to approximately 3.5 years)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 106 | 107
months | NA [NA to NA] — Median and corresponding CI could not be calculated due to low number of participants who had an event. | NA [NA to NA] — Median and corresponding CI could not be calculated due to low number of participants who had an event.

10. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) Questionnaire Visual Analogue Scale (VAS) Score
Description: EQ-5D VAS: participant rated questionnaire to assess health-related quality of life (QoL) in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, thereafter every 3 cycles from Cycle 3 to Cycle 45 (each cycle = 21 days)
Population: ITT population. Here, 'Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'n' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 102 | 102
units on a scale
  Baseline (n = 102, 102) | 69.7 (22.74) | 68.6 (23.58)
  Change at Cycle 3 (n = 83, 90) | 0.9 (19.31) | 1.7 (23.16)
  Change at Cycle 6 (n=68, 82) | 1.0 (23.59) | 4.3 (24.49)
  Change at Cycle 9 (n=67, 68) | 2.2 (23.00) | 6.6 (26.29)
  Change at Cycle 12 (n=53, 59) | -1.4 (30.19) | 6.8 (23.59)
  Change at Cycle 15 (n=43, 43) | 6.3 (19.34) | 8.1 (24.45)
  Change at Cycle 18 (n=32, 28) | 5.7 (21.83) | 6.5 (22.12)
  Change at Cycle 21 (n=30, 27) | 3.2 (20.00) | 1.3 (28.50)
  Change at Cycle 24 (n=25, 26) | 3.1 (17.06) | 2.8 (23.16)
  Change at Cycle 27 (n=21, 24) | 5.9 (18.79) | 1.1 (20.16)
  Change at Cycle 30 (n=18, 19) | 5.4 (19.87) | 9.5 (19.68)
  Change at Cycle 33 (n=15, 15) | 2.9 (24.03) | 13.4 (19.65)
  Change at Cycle 36 (n=14, 7) | 4.8 (17.37) | 7.3 (21.72)
  Change at Cycle 39 (n=6, 1) | 15.8 (19.85) | 50.0 (NA) — Standard deviation data was not available because only 1 participant was evaluable at indicated time point.
  Change at Cycle 42 (n=2, 0) | -5.0 (14.14) | NA (NA) — Data was not available because no participant was evaluable at indicated time point.
  Change at Cycle 45 (n=1, 0) | 5.0 (NA) — Standard deviation data was not available because only 1 participant was evaluable at indicated time point. | NA (NA) — Data was not available because no participant was evaluable at indicated time point.

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast (FACT-B) Questionnaire Score
Description: FACT-B questionnaire is used for assessment of health-related QoL in participants with breast cancer. It consists of 36 items, summarized to 5 subscales: physical (7 items), functional (7 items), social/family (7 items); all 3 ranged from 0 to 28, emotional (6 items) ranging from 0 to 24, and breast cancer subscale (9 items) ranging from 0 to 36; high subscale score represents a better QoL. All single-item measures ranges from 0='Not at all' to 4='Very much'. Total possible score ranged from 0 to 144. High scale score represents a better QoL.
Time Frame: Baseline, thereafter every 3 cycles from Cycle 3 to Cycle 45 (each cycle = 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Number analyzed (Participants) | 100 | 100
units on a scale
  Baseline (n = 100, 100) | 76.7 (13.46) | 78.5 (16.06)
  Change at Cycle 3 (n = 82, 90) | -1.96 (10.872) | -2.57 (13.159)
  Change at Cycle 6 (n=70, 79) | -0.97 (12.749) | 0.47 (13.724)
  Change at Cycle 9 (n=65, 60) | 1.44 (13.189) | -0.42 (14.602)
  Change at Cycle 12 (n=52, 51) | 0.40 (12.057) | 0.51 (14.510)
  Change at Cycle 15 (n=43, 44) | 2.72 (10.989) | 0.09 (13.713)
  Change at Cycle 18 (n=32, 32) | 4.58 (11.801) | 0.51 (16.512)
  Change at Cycle 21 (n=29, 24) | 3.22 (13.178) | -0.23 (16.116)
  Change at Cycle 24 (n= 26, 23) | 1.19 (10.660) | -1.03 (14.546)
  Change at Cycle 27 (n=20, 22) | 4.91 (9.900) | 0.55 (14.185)
  Change at Cycle 30 (n=18, 24) | 3.96 (11.082) | -0.26 (17.381)
  Change at Cycle 33 (n=14, 17) | 5.75 (13.272) | 1.76 (19.179)
  Change at Cycle 36 (n=15, 13) | 1.26 (9.210) | 2.74 (14.354)
  Change at Cycle 39 (n=6, 6) | -3.68 (16.866) | 7.33 (20.992)
  Change at Cycle 42 (n=4, 0) | -0.17 (10.599) | NA (NA) — Data was not available because no participant was evaluable at indicated time point.
  Change at Cycle 45 (n=1, 0) | 1.00 (NA) — Standard deviation data was not available because only 1 participant was evaluable at indicated time point. | NA (NA) — Data was not available because no participant was evaluable at indicated time point.

ADVERSE EVENTS:
Time Frame: Day 1 until 28 days after last study treatment (up to approximately 3.5 years)
Description: Treatment-emergent adverse events (TEAEs) are adverse events occurring between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. Safety Population included all participants who received at least one dose of any study treatment in any of the 2 cohorts.
Arm/Group | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion
Serious Adverse Events (participants affected / at risk) | 32/106 | 44/107
Other Adverse Events (participants affected / at risk) | 103/106 | 106/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion (N=106) | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion (N=107)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 6
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 5 | 0
Device related infection (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Sensorimotor disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab + Trastuzumab + Vinorelbine: Separate Infusion (N=106) | Pertuzumab + Trastuzumab + Vinorelbine: Single Infusion (N=107)
Anaemia (Blood and lymphatic system disorders) | 36 | 19
Leukopenia (Blood and lymphatic system disorders) | 24 | 16
Neutropenia (Blood and lymphatic system disorders) | 54 | 61
Tachycardia (Cardiac disorders) | 3 | 7
Cataract (Eye disorders) | 2 | 6
Lacrimation increased (Eye disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 15 | 19
Abdominal pain upper (Gastrointestinal disorders) | 20 | 22
Constipation (Gastrointestinal disorders) | 35 | 35
Diarrhoea (Gastrointestinal disorders) | 61 | 62
Dry mouth (Gastrointestinal disorders) | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 15
Haemorrhoids (Gastrointestinal disorders) | 9 | 4
Nausea (Gastrointestinal disorders) | 52 | 44
Stomatitis (Gastrointestinal disorders) | 19 | 26
Vomiting (Gastrointestinal disorders) | 34 | 25
Asthenia (General disorders) | 42 | 29
Chest pain (General disorders) | 7 | 10
Chills (General disorders) | 30 | 14
Extravasation (General disorders) | 1 | 7
Fatigue (General disorders) | 36 | 41
Influenza like illness (General disorders) | 7 | 9
Mucosal inflammation (General disorders) | 16 | 26
Oedema peripheral (General disorders) | 6 | 13
Pain (General disorders) | 7 | 12
Pyrexia (General disorders) | 35 | 22
Hypersensitivity (Immune system disorders) | 6 | 4
Conjunctivitis (Infections and infestations) | 8 | 3
Cystitis (Infections and infestations) | 8 | 16
Gastroenteritis (Infections and infestations) | 6 | 3
Influenza (Infections and infestations) | 11 | 4
Nasopharyngitis (Infections and infestations) | 20 | 15
Paronychia (Infections and infestations) | 2 | 6
Rhinitis (Infections and infestations) | 14 | 7
Sinusitis (Infections and infestations) | 4 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 15
Urinary tract infection (Infections and infestations) | 11 | 13
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 6
Alanine aminotransferase increased (Investigations) | 8 | 11
Aspartate aminotransferase increased (Investigations) | 4 | 10
Ejection fraction decreased (Investigations) | 9 | 2
Gamma-glutamyltransferase increased (Investigations) | 9 | 9
Weight decreased (Investigations) | 22 | 22
Weight increased (Investigations) | 1 | 6
Decreased appetite (Metabolism and nutrition disorders) | 23 | 24
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 28
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 29
Dizziness (Nervous system disorders) | 4 | 16
Dysgeusia (Nervous system disorders) | 9 | 8
Headache (Nervous system disorders) | 15 | 27
Neuropathy peripheral (Nervous system disorders) | 11 | 23
Paraesthesia (Nervous system disorders) | 20 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 10
Polyneuropathy (Nervous system disorders) | 5 | 8
Anxiety (Psychiatric disorders) | 2 | 10
Depression (Psychiatric disorders) | 10 | 8
Insomnia (Psychiatric disorders) | 10 | 19
Dysuria (Renal and urinary disorders) | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 21
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 12
Erythema (Skin and subcutaneous tissue disorders) | 9 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 6
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 9
Rash (Skin and subcutaneous tissue disorders) | 25 | 12
Hot flush (Vascular disorders) | 7 | 5
Hypertension (Vascular disorders) | 8 | 31
Hypotension (Vascular disorders) | 6 | 3
Phlebitis (Vascular disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.